CLINICAL TRIAL: NCT07003022
Title: An Open and Exploratory Phase Ⅱ Clinical Trial of Cadonilimab Combined With Anti-angiogenic Agents in Metastatic dMMR/MSI-H Colorectal Cancer
Brief Title: Phase Ⅱ Clinical Trial of Cadonilimab Combined With Anti-angiogenic Agents in Metastatic dMMR/MSI-H CRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBRC2025
Record Dates: First submitted 2025-06-02; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Colo-rectal Cancer; MSIhi or dMMR Advanced Unresectable or Metastatic Solid Tumors, Including Colorectal Cancers
MeSH Terms: conditions — Colonic Neoplasms | interventions — regorafenib; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immune-naive group (Experimental): Patients with no prior PD-1/PD-L1 treatment
  Interventions: Drug: cadonilimab combined with an anti-angiogenic agent, which is selected by the investigator from bevacizumab, regorafenib, or fruquintinib.
- Immune rechallenge group (Experimental): Patients who previously received and failed PD-1/PD-L1 therapy
  Interventions: Drug: cadonilimab combined with an anti-angiogenic agent, which is selected by the investigator from bevacizumab, regorafenib, or fruquintinib.

INTERVENTIONS:
Drug: cadonilimab combined with an anti-angiogenic agent, which is selected by the investigator from bevacizumab, regorafenib, or fruquintinib. — Cadonilimab: 10mg/kg Q3W; Bevacizumab: 7.5mg/kg Q3W; Regorafenib: 80mg QD; Fruquintinib: 3mg QD.

SUMMARY:
This study is a prospective, open-label, dual-arm exploratory Phase II clinical trial designed to assess the efficacy and safety of cadonilimab combined with anti-angiogenic agents in patients with dMMR/MSI-H recurrent or metastatic colorectal cancer. Eligible patients are enrolled into two cohorts based on their prior exposure to PD-1/PD-L1 antibody therapy: Cohort A (immune-naive group - patients with no prior PD-1/PD-L1 treatment) and Cohort B (immune rechallenge group - patients who previously received and failed PD-1/PD-L1 therapy). All participants receive combination therapy with cadonilimab and an anti-angiogenic agent, which is selected by the investigator from bevacizumab, regorafenib, or fruquintinib. Treatment continues until the occurrence of intolerable toxicity, disease progression, withdrawal of informed consent, loss to follow-up, death, other conditions deemed by the investigator to warrant discontinuation, or study termination-whichever occurs first. Cadonilimab treatment will not exceed two years. Tumor response is evaluated every six weeks using RECIST v1.1 criteria. Safety is assessed using CTCAE v5.0, and adverse events are recorded from the first dose to 30 days after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

- Signed written informed consent prior to enrollment. Age 18-80 years. dMMR or MSI-H Diagnosis confirmed by histological examination and/or cytological examination combined with imaging assessment of advanced colorectal cancer.

ECOG score: 0 to 2. At least one measurable lesion (≥10 mm long diameter on CT scan for non-lymph node lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to iRECIST criteria).

Adequate organ function with. Routine blood: Absolute Neutrophil Count (ANC) 1.5 × 109/L, Platelets (Platelet, PLT) ≥ 100 × 109/L, Hemoglobin (HGB) ≥ 90 g/L.

Liver function: Total Bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤3×ULN; serum albumin ≥30 g/L; after conventional hepatoprotective treatment meeting the above criteria, and can be stable for at least 1 week after evaluation by the investigator can be enrolled.

Renal function: Creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/mi (applying the standard Cockcroft-Gault formula).

Coagulation function: International Normalized Ratio (INR) ≤ 1.5 /PT ≤ 1.5 × ULN, aPTT ≤ 1.5 × ULN; if the subject is receiving anticoagulation therapy, as long as PT and INR are within the range drawn up by anticoagulant drugs.

A predicted survival of ≥ 3 months. Female patients must be non-pregnant and non-lactating and are required to use a medically approved form of contraception (e.g., IUD, pill or condom) during study treatment and for at least 120 days after study completion, and are not allowed to donate eggs to another person or freeze them for fertilization and propagation during this period.

Exclusion Criteria:

* Symptomatic brain metastases. A prior history of a primary tumor outside of the colorectal cancer in 3 years Active autoimmune disease or autoimmune disease with potential for recurrence such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery cannot be included; subjects with vitiligo or complete remission of asthma in childhood and adult who do not require any intervention afterwards can be included; subjects with asthma requiring medical intervention with bronchodilators cannot be included.

Subjects with any severe and/or uncontrolled disease. including. Poorly controlled blood pressure (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L) Having ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470ms) and ≥ grade 2 congestive heart failure (New York Heart Association [NYHA] classification) Active or uncontrolled severe infection (≥ CTCAE grade 2 infection) requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection Active hepatitis (transaminases do not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥ 1000 IU/ml or ≥ 10^4 copies/ml; hepatitis C reference: HCV RNA ≥ 1000 IU/ml or ≥ 10^4 copies/ml; after nucleotide based antiviral therapy below the above criteria, can be enrolled); chronic hepatitis B virus carriers with HBV DNA < 10^4 IU/ml, who must receive concomitant antiviral therapy during the trial to be enrolled.

Those with renal failure requiring hemodialysis or peritoneal dialysis. Those with a history of immunodeficiency, including HIV-positive or suffering from other acquired or congenital immunodeficiency diseases, or a history of organ transplantation Active autoimmune disease requiring systemic therapy (e.g., use of disease-relieving drugs, corticosteroids, or immunosuppressive agents) within 2 years prior to the start of study treatment, except for replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency); receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy. Doses >10 mg/day of prednisone or other equivalent hormone and within 2 weeks of the first dose and still continuing Those with a history of active tuberculosis Those who fail to control and still require repeated drainage of ascites, pericardial effusion, pleural effusion.

Research treatment related to. Patients who have undergone major organ transplantation Those who have undergone major surgical treatment, incisional biopsy or significant traumatic injury within 28 days prior to the start of study treatment; or have a long-standing untreated wound or fracture History of live attenuated vaccination within 14 days prior to the start of study treatment or planned live attenuated vaccination during the study History of severe hypersensitivity reactions following the use of monoclonal antibodies; known hypersensitivity to active ingredients or excipients such as envafolimab, lenvatinib, etc., of this study drug Those who are participating or have participated in other clinical studies within 4 weeks prior to the start of the study Those who have received PD-1/CTLA-4 dual immunotherapy during previous treatment.

Those with a history of severe allergy. Women who are pregnant or breastfeeding At risk for bleeding, or with coagulation disorders, or undergoing thrombolytic therapy Those with a history of psychotropic substance abuse and unable to abstain or with psychiatric disorders Subjects who, in the judgment of the investigator, have a concomitant disease that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or subjects for whom other reasons are deemed to exist that make them unsuitable for enrollment In the judgment of the investigator, subjects who, in the judgment of the investigator, have a concomitant disease that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or subjects for whom other reasons are deemed to exist that make them unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with measurable lesions achieving a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) criteria.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 12 months
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.
Disease Control Rate (DCR) | 12 months
  The proportion of participants who achieves a best overall response of CR, PR or stable disease(SD).
Duration of Response (DoR) | 12 months
  The time from the date that response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Overall Survival (OS) | 18 months
  OS is defined as the time from enrollment to death from any cause.
Adverse Events (AEs) | 12 months
  Adverse Events (AEs) according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No